CLINICAL TRIAL: NCT06967363
Title: Multi-modality Imaging and Collection of Biospecimen Samples in Understanding Brain Function in Low Back Pain Patients: a Longitudinal Cohort Study
Brief Title: Multimodal Imaging and Biospecimen Collection for Low Back Pain (LBPB)
Acronym: LBPB
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Jie Sun, associate professor, Peking University Third Hospital
Other Study IDs: M2023570
Record Dates: First submitted 2025-04-22; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Chronic Low Back Pain (CLBP); Acute Low Back Pain; Low Back Pain; Chronic Pain; Acute Pain; Mental Disorders; Sleep Disorder; Fibromyalgia (FM); Nociplastic Pain; Neuropathic Pain; Nonspecific Low Back Pain
Keywords: chronic low pack pain; fMRI; brain function; microbiota; nociplastic pain; treatment
MeSH Terms: conditions — Low Back Pain; Chronic Pain; Acute Pain; Mental Disorders; Sleep Wake Disorders; Fibromyalgia; Nociplastic Pain; Neuralgia | interventions — Nerve Block; Dosage Forms; Celecoxib; Ibuprofen; Diclofenac; Pregabalin; Etoricoxib; loxoprofen; Psychotherapy; Cognitive Behavioral Therapy; Acceptance and Commitment Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood; Faces
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-surgical group: Participants receiving conventional treatment such as medication , exercise, physical therapy, psychotherapy ( acceptance and realization therapy, pain reprocessing therapy, and cognitive behavior therapy) etc.,
  Interventions: Drug: Medication; Behavioral: Psychotherapy
- Surgical group: Participants undergoing surgical interventions, such as nerve block, or endoscopic lumbar discectomy.
  Interventions: Procedure: Nerve Block; Procedure: endoscopic spinal disecetomy

INTERVENTIONS:
Procedure: Nerve Block — The "nerve block" intervention in this study involves the targeted administration of anesthetic agents and corticosteroids to specific nerves or nerve roots to alleviate pain associated with low back pain. This procedure is performed under imaging guidance (e.g., fluoroscopy or ultrasound) to ensure precise delivery of the medication to the affected nerve. It aims to temporarily block the transmission of pain signals from the affected area to the brain, providing relief and allowing for a better assessment of the underlying pain mechanism. The nerve block is distinguished from other interventions in this study by its localized approach, focusing on pain modulation through direct neural targeting, rather than systemic pain management methods. The procedure may be used either as a standalone treatment or in conjunction with other therapies (e.g., physical therapy, medications) based on the patient's individual needs and response to treatment.
  Other Names: Selective Nerve Root Block (SNRB); Transforaminal Epidural Injection
  Groups: Surgical group
Procedure: endoscopic spinal disecetomy — The Endoscopic Lumbar Discectomy is a minimally invasive surgical procedure designed to treat symptomatic lumbar disc herniations by removing the protruding or damaged disc material that is pressing on the nerve roots. This intervention is distinguished by the use of endoscopic technology, which allows for a smaller incision, real-time visualization of the affected area via an endoscope, and the removal of herniated disc tissue with minimal disruption to surrounding structures. Unlike traditional open discectomy, which requires larger incisions and muscle dissection, endoscopic discectomy involves the use of a small tubular retractor and specialized instruments, leading to reduced blood loss, shorter recovery times, and less postoperative pain.
  This procedure is typically performed under local anesthesia, and the patient is often able to go home the same day. It is specifically designed for patients with lumbar disc herniations who have not responded to conservative way.
  Other Names: endoscopic lumbar disecetomy; Endoscopic Discectomy; Percutaneous Endoscopic Lumbar Discectomy
  Groups: Surgical group
Drug: Medication — The treatment of lumbar pain typically involves a multimodal approach combining medications based on the specific type of pain and patient needs. NSAIDs, acetaminophen, and muscle relaxants are often first-line treatments for nociceptive pain, while opioids and anticonvulsants like pregabalin are used for more severe or neuropathic pain. The choice of medication is guided by the severity of the pain, its underlying causes, and the patient's response to treatment. Each class of medication has its strengths and limitations, and the decision to use them must take into account factors like patient safety, the risk of side effects, and long-term efficacy.
  Other Names: celecoxib; ibuprofen; diclofenac; Pregabalin; Lyrica; Etoricoxib; loxoprofen
  Groups: Non-surgical group
Behavioral: Psychotherapy — Cognitive Behavioral Therapy (CBT): This structured, goal-oriented therapy focuses on identifying and changing negative thought patterns, cognitive distortions, and maladaptive behaviors associated with chronic pain. CBT equips patients with coping strategies to reframe thoughts, reduce pain-related anxiety, and enhance emotional regulation, thereby improving overall function and quality of life. CBT can include techniques such as cognitive restructuring, relaxation training, and behavioral activation.
  Acceptance and Commitment Therapy (ACT): ACT encourages individuals to accept pain and distressing emotions rather than avoiding them. It emphasizes mindfulness, acceptance, and values-based living, helping patients focus on behaviors that align with their values, despite ongoing pain.
  Other Names: cognitive behavioral therapy; Acceptance and Commitment Therapy
  Groups: Non-surgical group

SUMMARY:
This prospective cohort study investigates the neurobiological, genetic, and psychosocial mechanisms underlying acute and chronic low back pain (LBP). Core objectives include establishing a high-quality biobank to support future research in connectomics, genomics, and biomarker discovery, and identifying predictors of pain progression and treatment response.

The study will also assess the impact of comorbid conditions such as anxiety, depression, and sleep disturbances on pain perception and clinical outcomes. Longitudinal analyses will explore the dynamic interplay between emotion, cognition, sleep, and pain to inform precision, mechanism-based interventions.

Functional imaging will be used to examine brain responses to nociceptive modulation, aiming to identify neural circuits involved in pain chronification. By integrating multimodal data-including neuroimaging, neurophysiology, microbiota profiling, polysomnography, and molecular assays-the study will define LBP subtypes, with a particular focus on nociceptive, neuropathic, and nociplastic mechanisms. The ultimate goal is to establish prognostic biomarkers and advance personalized strategies for LBP prevention and treatment.

DETAILED DESCRIPTION:
Low back pain (LBP) is one of the leading causes of disability globally, yet its underlying mechanisms remain poorly understood. Clinical management is often challenging due to the heterogeneity in symptom presentation and treatment response. Current approaches range from self-management and pharmacological therapies to targeted interventions, including nerve blocks and surgery. To address these challenges, this prospective, longitudinal cohort study is designed to comprehensively investigate the neurobiological, genetic, microbiological, and psychosocial factors contributing to the onset, maintenance, and variability of LBP.

The study includes individuals with both acute and chronic LBP to capture diverse clinical trajectories and identify determinants of recovery versus chronification. A central objective is to establish a well-curated biobank containing high-quality biospecimens (e.g., blood, stool) and multimodal datasets to facilitate future research in genomics, connectomics, microbiome science, and biomarker discovery.

Following a one-week run-in period to confirm eligibility, participants undergo comprehensive, multidimensional phenotyping. This includes clinical evaluation, self-reported outcomes, quantitative sensory testing, polysomnography (PSG), structural and functional magnetic resonance imaging (fMRI), heart rate variability (HRV), and microbiota profiling. Treatments-including conservative care (e.g., medications, health education), interventional procedures (e.g., nerve blocks), or surgery (e.g., endoscopic lumbar discectomy)- will be administered based on individualized clinical assessment.

All participants will undergo deep phenotyping at baseline, with follow-up assessments at 1 month, 3 months, 6 months and 1 year post-enrollment. Functional MRI scans will be conducted at baseline; 1 day before and after surgery or interventional procedures (if applicable); and at 1 month, 3 months, 6 months, and 1 year. If patients do not show significant improvement within 4 weeks or experience worsening symptoms, their treatment will be reassessed, and secondary interventions such as CBT, alternative medications, or further surgery will be considered based on their needs and progress.

The study investigates key systems involved in pain processing and chronification, including brain networks, central and peripheral nervous system activity, immune and inflammatory pathways, autonomic regulation, and the gut-brain axis. Longitudinal tracking will be used to analyze changes in these biological systems and their associations with clinical outcomes such as pain persistence, sleep quality, emotional distress, and functional status. Ultimately, this research aims to identify mechanistic biomarkers and define LBP subtypes to support the development of personalized, mechanism-based interventions for more effective prevention and treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 to 80 years.
2. Diagnosis of low back pain, defined as pain located between the lower costal margins and the gluteal folds, with or without leg pain.
3. Eligible for surgical or non-surgical treatments.
4. Willingness to undergo neuroimaging (fMRI), microbiota sampling, psychological assessments, and other related study procedures. Ability to provide written informed consent.

Exclusion Criteria:

1. Severe neurological deficits requiring emergency surgery.
2. Antibiotic or probiotic use within the past 4 weeks. Suffering from digestive diseases such as irritable bowel syndrome, gastric ulcer, duodenal ulcer, etc.;
3. Diagnosed spinal infections, tumors, fractures, or inflammatory diseases (e.g., ankylosing spondylitis).
4. Known severe psychiatric disorders (e.g., schizophrenia, bipolar disorder) that would interfere with study participation.Head trauma; history of substance abuse.
5. Contraindications to MRI scanning (e.g., pacemaker, metallic implants, severe claustrophobia).
6. Pregnant or breastfeeding women.
7. Participation in another interventional clinical trial within the past 3 months.
8. Working at night shifts or travelling across time zones in the past 6 months.
9. Excessive consumption of coffee, tea.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Peking University Third Hospital
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity (Brief Pain Inventory - Short Form) | Baseline; 1 week after treatment; 2 weeks after treatment; 1 month after treatment; 3 months after treatment; 6 months after treatment; 12 months after treatment
  Pain intensity will be assessed using the BPI-SF pain severity subscale, consisting of four 0-10 numeric ratings: worst, least, average, and current pain over the past 24 hours. The primary outcome will be the average of these four items. Higher scores indicate greater pain severity.
Pain Interference (Brief Pain Inventory - Short Form) | Time Frame: Baseline; 1 week after treatment; 2 weeks after treatment; 1 month after treatment; 3 months after treatment; 6 months after treatment; 12 months after treatment
  Pain interference will be measured using the BPI-SF interference subscale, which includes seven items assessing interference with general activity, mood, walking ability, normal work, relations with others, sleep, and enjoyment of life. Each item is scored on a scale of 0 (does not interfere) to 10 (completely interferes). The mean of the seven items will be reported as the interference score.

SECONDARY OUTCOMES:
Pain Catastrophizing Scale (PCS) | Time Frame: Baseline; 1 week after treatment; 2 weeks after treatment; 1 month after treatment; 3 months after treatment; 6 months after treatment; 12 months after treatment
  The PCS consists of 13 items, each rated on a 0 (not at all) to 4 (all the time) scale. Total scores range from 0 to 52, with higher scores indicating greater pain catastrophizing. The total PCS score will be used as the outcome.
Pain Coping Strategies Questionnaire | Baseline; 2 weeks after treatment; 1 month after treatment; 3 months after treatment; 6 months after treatment; 12 months after treatment
  Use of this scale is designed to measure psychological and behavioral strategies for how individuals cope with chronic pain. Participants need to rate each item on a scale of 0 (never) to 6 (always), depending on the situation.
Pain Resilience Scale | Baseline; 2 weeks after treatment; 1 month after treatment; 3 months after treatment; 6 months after treatment; 12 months after treatment
  This scale is used to assess an individual's mental resilience in response to pain, including the capacity of adaptive, cognitive, affective, and behavioral strategies during the pain experience. Participants need to rate each item on a scale of 0 (never) to 4 (always), depending on the situation.
Pain Self-efficacy Scale | Baseline; 2 weeks after treatment; 1 month after treatment; 3 months after treatment; 6 months after treatment; 12 months after treatment
  This scale is used to assess an individual's confidence in managing pain, with higher scores indicating greater confidence in pain management. Participants need to rate each item on a scale of 0 (never) to 6 (always), depending on the situation.
Central Sensitization Scale | Baseline; 2 weeks after treatment; 1 month after treatment; 3 months after treatment; 6 months after treatment; 12 months after treatment
  This scale is used to comprehensively assess an individual's level of central sensitization, with higher scores indicating a higher level of central sensitization and greater sensitivity to painful stimuli. Participants need to rate each item on a scale of 0 (never) to 4 (always), depending on the situation.
Brief Family Relationships Scale | Baseline
  This scale is used to assess the quality of family relationships and provides insight into the interaction, support, communication, and conflict among family members. Participants need to rate each item on a scale of 0 (Strongly agree) to 6 (Strongly disagree), depending on the situation.
Family Pain Questionnaire | Baseline
  The scale contains 16 questions about pain and pain relief, and each question needs to be scored on a scale of approval, with a scale of 0 to 10 indicating an increase in degree, with higher scores representing greater agreement with the statement.
Dietary Patterns (Structured Dietary Questionnaire - Food Frequency Component) | Baseline
  Dietary patterns will be assessed using a structured dietary questionnaire that includes a food frequency component. Participants report the frequency of consumption of various food groups (e.g., fruits, vegetables, dairy, meats, processed foods) over a defined period. Data will be used to calculate dietary diversity and adherence scores. There is no single summary score; results are used descriptively and for correlation analyses.
Sensory Threshold and Pain Perception as Assessed by Quantitative Sensory Testing (QST) Using Mechanical and Electrical Stimulation | Baseline; 1 day after treatment; 1 month after treatment; 3 months after treatment; 6 months after treatment; 12 months after treatment
  Sensory gain or loss will be assessed using Quantitative Sensory Testing (QST) through both mechanical and electrical stimuli applied to multiple body sites (left leg, right leg, lumbar region, left arm, right arm).
  Mechanical stimulation will be delivered using Von Frey filaments (0.008g to 300g). The mechanical detection threshold will be recorded in grams. Lower values indicate greater tactile sensitivity.
  Electrical stimulation will be administered using surface electrodes with adjustable intensity (0-110 volts). The electrical pain threshold will be recorded in volts. Higher voltage indicates a higher pain threshold.
  Participants will also provide subjective ratings of pain unpleasantness on a Numeric Rating Scale from 0 (no unpleasantness) to 10 (most unpleasant imaginable).
Quantitative Sensory Testing (Electrical stimulation) | Baseline; 1 day after treatment; 2 weeks after treatment; 1 month after treatment; 3 months after treatment; 6 months after treatment; 12 months after treatment
  An electrical stimulation device (STM200) will be used to administer a series of electrical stimulation of different intensities (voltage range 0-100V) to record the sensations corresponding to the different stimulation intensities. The lower the value, the more sensitive the perception.
Oswestry Disability Index | Baseline; 2 weeks after treatment; 1 month after treatment; 3 months after treatment; 6 months after treatment; 12 months after treatment
  The Oswestry Disability Index (ODI) is a validated, self-reported questionnaire used to assess functional disability related to low back pain. It consists of 10 sections measuring limitations in activities such as pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life, social life, and traveling.
  Each section is scored from 0 to 5, resulting in a total score ranging from 0 to 50, which is then converted to a percentage (0%-100%). Higher scores indicate greater disability.
Health-Related Quality of Life as Assessed by the 36-Item Short Form Health Survey (SF-36) | Baseline; 1 month after treatment; 3 months after treatment; 6 months after treatment; 12 months after treatment
  The SF-36 is a validated, self-administered questionnaire that evaluates health-related quality of life across 8 domains: physical functioning, role limitations due to physical health, role limitations due to emotional problems, vitality, emotional well-being, social functioning, bodily pain, and general health perceptions.
  Scores for each domain range from 0 to 100, with higher scores indicating better health status or functioning. The survey can also be summarized into two component scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS), both scaled from 0 to 100.
Pittsburgh Sleep Quality Index | Baseline; 1 month after treatment; 3 months after treatment; 6 months after treatment; 12 months after treatment
  This scale mainly assesses subjective sleep in the past month, including sleep duration, sleep efficiency, sleep medication use, and sleep disorders. The total score ranges from 0-21, with higher scores indicating worse sleep quality.
Polysomnography | Baseline; 1 day after treament; 1 month after treatment; 3 months after treatment; 6 months after treatment; 12 months after treatment
  Polysomnography, a device produced by Compumedics, is used to record and analyze physiological indicators of the human body during sleep, including electroencephalography, electrocardiography, electromyography, electrooculography, oral and nasal airflow, blood oxygen saturation, leg movement, right leg movement, pulse rate, etc.
Insomnia Severity Index | Baseline; 2 weeks after treatment; 1 month after treatment; 3 months after treatment; 6 months after treatment; 12 months after treatment
  This scale is used to assess the severity of insomnia symptoms in the past two weeks, including difficulty falling asleep, difficulty maintaining sleep, early waking, and concern about sleep problems. The higher the score, the more serious the insomnia symptoms.
Hamilton Anxiety Scale | Baseline; 2 weeks after treatment; 1 month after treatment; 3 months after treatment; 6 months after treatment; 12 months after treatment
  The Hamilton Anxiety Rating Scale (HAM-A) is a clinician-administered assessment used to measure the severity of a patient's anxiety. It includes 14 items, each assessing a symptom of anxiety (e.g., tension, fears, insomnia, somatic complaints).
  Each item is scored on a scale from 0 (not present) to 4 (severe), producing a total score ranging from 0 to 56. Higher scores indicate more severe anxiety. Scores can be interpreted as:
  0-17: mild severity
  18-24: mild to moderate severity
  25-30: moderate to severe
Hamilton Depression Scale | Baseline; 2 weeks after treatment; 1 month after treatment; 3 months after treatment; 6 months after treatment; 12 months after treatment
  This scale is used to assess the severity of depressive symptoms. The total score is between 0 and 63. The higher the score, the more severe the depression.
Patient Health Questionnaire-9 | Baseline; 2 weeks after treatment; 1 month after treatment; 3 months after treatment; 6 months after treatment; 12 months after treatment
  This scale is used to self-assess the severity of depressive symptoms. The total score is between 0 and 27. The higher the score, the more severe the depression.
Generalized Anxiety Disorder Scale-7 | Baseline; 2 weeks after treatment; 1 month after treatment; 3 months after treatment; 6 months after treatment; 12 months after treatment
  This scale is used to self-assess the severity of anxiety symptoms. The total score is between 0 and 21. The higher the score, the more severe the anxiety.
UCLA Loneliness Scale | Baseline; 2 weeks after treatment; 1 month after treatment; 3 months after treatment; 6 months after treatment; 12 months after treatment
  This scale is used to assess an individual's feelings of loneliness. Higher scores indicate greater loneliness.
Trail Making Test | Baseline; 3 months after treatment; 6 months after treatment; 12 months after treatment
  This test consists of 2 parts to assess executive function, attention and processing speed. TMT-A is to make a trail in numerical order; TMT-B is to make a trail from small to large alternating numbers and letters.
Stroop Test | Baseline; 3 months after treatment; 6 months after treatment; 12 months after treatment
  This test consists of four colors, "red, blue, yellow, and green," and requires that the meaning of the words be ignored and that choices be made based on the color. It is designed to assess cognitive inhibition and executive function.
Attention Network Test | Baseline; 3 months after treatment; 6 months after treatment; 12 months after treatment
  This test assesses executive functioning, vigilance, orientation, and other abilities by calculating the choice of arrow direction under different conditions.
Mnemonic Similarity Task | Baseline; 3 months after treatment; 6 months after treatment; 12 months after treatment
  This test determines hippocampal functioning by learning a series of images and then categorizing the images, including old images (exactly the same as those that have appeared before); new images (not at all the same as those that have appeared before); and similar images (similar to those that have appeared before but with differences).
Cognitive Flexibility Task | Baseline; 3 months after treatment; 6 months after treatment; 12 months after treatment
  This test determines cognitive flexibility by choosing the correct figure out of two patterns where the correct answer is reversed after a certain pattern.
Pain Empathy Task | Baseline; 3 months after treatment; 6 months after treatment; 12 months after treatment
  This task focuses on an individual's ability to perceive and understand pain in others and the relationship between pain empathy and the experience of pain in the self.
Pain Think/No-Think | Baseline; 3 months after treatment; 6 months after treatment; 12 months after treatment
  This task is mainly used to study how individuals actively control pain memory and pain experience.
Microbiota Analysis | Baseline; 3 months after treatment; 6 months after treatment; 12 months after treatment
  Fecal specimens will be collected, frozen, and centralized for analysis such as macro-genome sequencing.
Blood Sample Analysis | Baseline; 3 months after treatment; 6 months after treatment; 12 months after treatment
  Whole blood will be collected, centrifuged to separate plasma and blood cells, and centralized for analysis of inflammatory factors (IL-1β, TNF-α, IL-6, IL-10, TGF-β, etc), high-throughput gene sequencing.
Sleep Diary | Baseline; 1 day after treatment; 2 weeks after treatment; 1 month after treatment; 3 months after treatment; 6 months after treatment; 12 months after treatment
  The scale will be used to record subjective sleep. Participants actively reported the time to go to bed, time to wake up, sleep medication use, dim or bright sleep environment, and mental state after waking up.
MRI Scan | Baseline; 1 day after treatment; 1 month after treatment; 3 months after treatment; 6 months after treatment; 12 months after treatment
  The MRI scan includes structural imaging (lumbar and head) and functional imaging (Pain Sensitivity Task, Pain Empathy Task, Pain Think/No-Think, Mnemonic Similarity Task, Cognitive Flexibility Task, etc.).
Heart Rate Variability | Baseline; 1 day after treatment; 2 weeks after treatment; 1 month after treatment; 3 months after treatment; 6 months after treatment; 12 months after treatment
  The method is used to record changes in the time interval of the heartbeat, reflecting the degree to which the heart is regulated by the autonomic nervous system.
Adverse Event Record | Baseline; 2 weeks after treatment; 1 month after treatment; 3 months after treatment; 6 months after treatment; 12 months after treatment
  This scale is used to record whether adverse reactions such as fever, wound infection, vascular/neurologic injury, headache, fatigue, lower extremity swelling occurred.
Pain Sensitivity Scale | Baseline; 2 weeks after treatment; 1 month after treatment; 3 months after treatment; 6 months after treatment; 12 months after treatment
  This scale is used to access the degree of sensitivity to pain. Participants will be given different scenarios and access the most compatible pain intensity on a scale of 0-10.
Somatization Symptoms disorder-12 | Baseline; 2 weeks after treatment; 1 month after treatment; 3 months after treatment; 6 months after treatment; 12 months after treatment
  This scale is a tool used to assess whether an individual experiences somatization symptoms.
Chronic Pain Helplessness Scale | Baseline; 2 weeks after treatment; 1 month after treatment; 3 months after treatment; 6 months after treatment; 12 months after treatment
  This scale is used to assess the participant's feelings of helplessness regarding chronic pain. Participants need to rate each item on a scale of 0 (strongly disagree) to 5 (strongly agree), depending on the situation.
Thought Control Scale | Baseline; 2 weeks after treatment; 1 month after treatment; 3 months after treatment; 6 months after treatment; 12 months after treatment
  This scale is used to assess an individual's ability to control their thinking in response to negative emotions or stress.
Pain Empathy Scale | Baseline; 2 weeks after treatment; 1 month after treatment; 3 months after treatment; 6 months after treatment; 12 months after treatment
  This scale is used to assess an individual's ability to empathize with others in pain.
Complete Blood Count | Baseline
  Routine blood count is a test that measures the number and proportion of various cells in our blood, mainly including the number and proportion of red blood cells, white blood cells and platelets.
Family Depression and Anxiety Scores (PHQ-9 and GAD-7) | Baseline
  Depression will be assessed using the Patient Health Questionnaire-9 (PHQ-9), with scores ranging from 0 to 27. Anxiety will be assessed using the Generalized Anxiety Disorder-7 (GAD-7) scale, with scores ranging from 0 to 21. Higher scores reflect greater symptom severity.
Family Sleep Quality Score (Pittsburgh Sleep Quality Index - PSQI) | Baseline
  The PSQI is a self-rated questionnaire that assesses sleep quality over the past month. It yields a global score ranging from 0 to 21, with higher scores indicating poorer sleep quality.
Family Functioning Score (Brief Family Relationship Scale) | Baseline
  Family functioning will be assessed using the Brief Family Relationship Scale, which evaluates cohesion, expressiveness, and conflict. Each subscale is scored separately; higher cohesion and expressiveness scores and lower conflict scores indicate healthier family dynamics.
Age | Baseline
  Participant's age will be collected at baseline as a continuous variable in years.
Gender (Male/Female/Other) | Baseline
  Participant's gender identity will be recorded at baseline.
Height (cm) | Baseline
  Participant's height measured in centimeters.
Weight (kg) | Baseline
  Participant's weight measured in kilograms.
Ethnicity (Self-Reported) | Baseline
  Participant's self-identified ethnicity will be recorded at baseline using predefined categories.
Education Level | Baseline
  Education level will be self-reported using predefined categories (e.g., high school, college, graduate).
Employment Status | Baseline
  Current employment status will be recorded at baseline.
Marital Status | Baseline
  Marital status will be collected at baseline (e.g., single, married, divorced).
Smoking History | Baseline
  Smoking history will be collected at baseline, including current smoking status and past use.
Alcohol Consumption | Baseline
  Alcohol consumption history will be collected at baseline (e.g., frequency and amount).
Medical History | Baseline
  Medical history including relevant comorbidities will be collected at baseline via participant self-report and medical record review.
Blood Biochemistry | Baseline
  This item evaluates liver function, renal function, etc. by examining venous blood. The main test items include: alanine aminotransferase, creatinine, urea nitrogen, serum glucose, triglyceride, total cholesterol.
Electromyography | Baseline
  By recording the electrical activity of muscles and nerves, muscle function and peripheral nervous system abnormalities are evaluated.
Income | Baseline
  Collect the range of participants' monthly income, in RMB, for example: no income, 1-999, 1000-1999, 2000-3999, 4000-5999, 6000-7999, 8000-9999, 10000-14999, 15000-19999, 20000-24999, 25000-39999, more than 40000.
Eating Habits (Structured Dietary Questionnaire - Behavioral Component) | baseline
  Eating habits, including meal frequency, snacking behavior, eating speed, and time of day of food consumption, will be assessed via a behavioral component of the structured dietary questionnaire. Responses are categorical or ordinal, used for descriptive and exploratory correlation analyses without a total score.
Bowel Habits (Structured Dietary Questionnaire - Bowel Function Component) | baseline
  Bowel habits will be evaluated using items in the dietary questionnaire that assess bowel movement frequency, stool consistency (e.g., via Bristol Stool Form Scale), and presence of gastrointestinal symptoms. Data are collected as categorical variables and will be used descriptively or to correlate with other outcomes (e.g., microbiome profile).

CONTACTS AND LOCATIONS:
Overall Officials: Jie Sun, Principal Investigator — Peking University Third Hospital
Locations (2):
- China (2):
  - Peking university third hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) that underlie the results reported in the published articles, after de-identification, will be shared. This includes demographic information, primary and secondary outcome measures, and relevant baseline characteristics. Data will be made available upon reasonable request for academic purposes, following institutional data-sharing policies and ethics approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Individual Participant Data (IPD) and supporting information will be made available starting from the publication date of the study results. The data will be accessible for a period of 5 years, from December 2025 to December 2030. During this period, the data will be available upon reasonable request for academic purposes, in accordance with the institutional data-sharing policies.
Access Criteria: Only approved researchers from academic institutions, research organizations, and government agencies who have a legitimate academic research purpose will be eligible to access the data. All individuals requesting access must adhere to the data use agreement and ensure the data will be used exclusively for research purposes.
  Authorized researchers will have access to de-identified individual participant data (IPD), which includes:
  Participant demographic information Primary and secondary outcome measures such as pain assessments, sleep quality, and neuroimaging data Study protocol, statistical analysis plan (SAP), and clinical study report (CSR) Informed consent form templates and ethics committee approval documents
  Data and supporting information will be made available through the official data-sharing platform of the research institution.
URL: https://www.pku.edu.cn